CLINICAL TRIAL: NCT05857020
Title: Battlefield Auricular Acupressure (BAApress) for Chronic Pain Management in Patients With Interstitial Cystitis/Bladder Pain Syndrome (IC/BPS)
Brief Title: Auricular Acupressure Therapy for Patients With IC/BPS
Acronym: IC/BPS
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: withdrawn by the sponsor due to personal constraints and limited funding
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00090489
Record Dates: First submitted 2023-04-18; First posted 2023-05-12 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-04

CONDITIONS: Interstitial Cystitis; Bladder Pain Syndrome; Urologic Diseases; Chronic Pain
Keywords: interstitial cystitis; bladder pain syndrome; pelvic pain; urologic pain; urologic disease
MeSH Terms: conditions — Cystitis, Interstitial; Urologic Diseases; Chronic Pain; Pelvic Pain

STUDY DESIGN:
Intervention Model Description: Any patient who has been scheduled for a provider visit in the Urology clinic for a diagnosis of interstitial cystitis/bladder pain syndrome (IC/BPS) who fulfills eligibility criteria will be considered for participation in this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Auricular Acupressure (AA) Group (Experimental): Participants will receive the AA intervention over a 5 day period in addition to their Standard of Care treatment for Interstitial Cystitis/Bladder Pain Syndrome (IC/BPS), and complete daily study questionnaires
  Interventions: Device: Auricular Acupressure

INTERVENTIONS:
Device: Auricular Acupressure — Auricular Acupressure (AA) utilizing all-natural vaccaria ear seeds will be applied to 5 designated sites on each participant's ear (total of 10 seeds placed per patient).
  Participants will be asked if they consent to having their ear placement photographed after placement (optional) and audio recorded during interventionist ear seed placement (optional) in collaboration with the BAApress training fidelity study.

SUMMARY:
The purpose of this study is to determine the feasibility of administering auricular acupressure for patients with interstitial cystitis/bladder pain syndrome (IC/BPS), and evaluating the efficacy of auricular acupressure to reduce pain scores and decrease pain medication usage over time.

DETAILED DESCRIPTION:
Eligible participants will be asked to complete baseline questionnaires. After completion, a study interventionist will place 10 adhesive acupressure pads/seeds on the participant's ears (5 on each ear). Each seed will be placed on a specific site on the ear believed to help with pain and overall well-being. Over the course of 5 days, participants will be asked to apply a small amount of manual pressure with their fingers to each of the ear pads and answer daily study questionnaires.

This feasibility trial is being conducted in collaboration with the Battlefield Auricular Acupressure (BAApress) Training and Intervention Fidelity study (IRB00084011).

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* History of documented interstitial cystitis/bladder pain syndrome (IC/BPS)
* Able to read and understand informed consent form in English

Exclusion Criteria:

* Patients with a history of skin disease (e.g. psoriasis) involving the ear, adhesive allergy, recent scar tissue on ear, or current abrasions or cuts on the ear
* Cognitive impairment (e.g. delirium, dementia)
* Physical impairment preventing them from applying daily pressure/stimulation to ear seeds
* Patients with cardiac pacemakers (contraindication to POINTER PAL)
* Use of some types of hearing aids (which could potentially obstruct placements of ear seeds)
* Any acute illness or psychiatric conditions that would impact adherence to the study requirements

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-07 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Pain scores using Numeric Rating Scale (NRS) | Baseline
  The NRS pain score is an 11-point pain scale in which patients will be asked to circle a number between 0 and 10 that best represents their current pain intensity. 0 usually indicates "no pain at all" and 10 indicates "worst pain imaginable."
Pain scores using Numeric Rating Scale (NRS) | Day 1
  The NRS pain score is an 11-point pain scale in which patients will be asked to circle a number between 0 and 10 that best represents their current pain intensity. 0 usually indicates "no pain at all" and 10 indicates "worst pain imaginable."
Pain scores using Numeric Rating Scale (NRS) | Day 2
  The NRS pain score is an 11-point pain scale in which patients will be asked to circle a number between 0 and 10 that best represents their current pain intensity. 0 usually indicates "no pain at all" and 10 indicates "worst pain imaginable."
Pain scores using Numeric Rating Scale (NRS) | Day 3
  The NRS pain score is an 11-point pain scale in which patients will be asked to circle a number between 0 and 10 that best represents their current pain intensity. 0 usually indicates "no pain at all" and 10 indicates "worst pain imaginable."
Pain scores using Numeric Rating Scale (NRS) | Day 4
  The NRS pain score is an 11-point pain scale in which patients will be asked to circle a number between 0 and 10 that best represents their current pain intensity. 0 usually indicates "no pain at all" and 10 indicates "worst pain imaginable."
Pain scores using Numeric Rating Scale (NRS) | Day 5
  The NRS pain score is an 11-point pain scale in which patients will be asked to circle a number between 0 and 10 that best represents their current pain intensity. 0 usually indicates "no pain at all" and 10 indicates "worst pain imaginable."
Change in Pain, Enjoyment, and General Activity (PEG) Assessment Scores | Day 5
  The PEG assesses a patient's reported intensity of pain and interference with general activity. It involves three 11-point numeric rating scales (NRS) ranging from 0 ("no pain" or "does not interfere") to 10 ("pain as bad as you can imagine" or "completely interferes"). Scores from each NRS will be compared before and after use of the study intervention. Higher scores represent more pain and or increased enjoyment and activity interference.

SECONDARY OUTCOMES:
Change in amount of Opioid Use | Baseline, Day 1, Day 2, Day 3, Day 4, Day 5
  Participants will be required to document all medications used prior to initiating therapy, and document all medications used while using the auricular acupressure seeds. Information collected will include medication type, frequency of use, and amount (milligrams) used. Mean/median changes from baseline to Day 5 will be calculated.
Pain Catastrophizing Scale (PCS) Assessments | Baseline and Day 5
  The PCS assesses the extend of catastrophic thinking due to pelvic/bladder pain according to 3 components: rumination, magnification, and helplessness. It is a 13-item scale with a total score range from 0 to 52. Each individual question is aimed to assess the thoughts and feelings of the patient using questions that are rated from 0 (not at all) to 4 (all the time). Higher scores are associated with higher amounts of pain catastrophizing.
Auricular Acupressure Acceptability - Likert scale scores | Day 5
  Participants will be asked 3 different questions to evaluate overall acceptance of the intervention (auricular acupressure). Responses will be analyzed quantitatively and qualitatively.
  1) The Likert scale question will be phrased as, "How satisfied were you with how your pain has been treated?" with the scale responses ranging from "5 = Very satisfied, 4 = Satisfied, 3 = Somewhat satisfied, 2 = Somewhat dissatisfied, 1 = Dissatisfied, 0 = Very dissatisfied."
Auricular Acupressure Acceptability - auricular acupressure | Day 5
  Participants will be asked 3 different questions to evaluate overall acceptance of the intervention (auricular acupressure). Responses will be analyzed quantitatively and qualitatively.
  2) The Yes/No question will be phrased as, "Would you consider using auricular acupressure in the future for pain or if recommended by your nurse of physician?" with responses ranging from "No, I would not use again" (score = 0), "Maybe" (score = 1), and "Yes, I would consider using it in the future" (Score = 2).
Auricular Acupressure Acceptability - Feedback | Day 5
  Participants will be asked 3 different questions to evaluate overall acceptance of the intervention (auricular acupressure). Responses will be analyzed quantitatively and qualitatively.
  3) The open-ended question will ask, "Is there anything else you would like to tell us that may be helpful for us to know regarding ear acupressure?" Each answer will be collected and assessed for future studies.
Change in Patient Global Impression of Change (PGIC) | Day 5
  The PGIC is a patient-reported assessment of improvement or decline in regard to their pain using a 7-point scale. Responses range from (1) "no change (or condition has got worse)" to (7) "a great deal better, and a considerable improvement that has made all the difference." This questionnaire also includes an 11-point NRS scale asking patient's to circle the number from 0 (much better) to 10 (much worse) that best describes the degree of change experienced since beginning the intervention.
Change in Patient-Reported Outcomes Measurement Information System (PROMIS) Sleep Disturbance Short Form | Baseline and Day 5
  This PROMIS sleep disturbance short form aims to assess a patient's reported quality of sleep. Each of the 6 items in the questionnaire is rated on a 5-point scale ranging from 1 (very good) to 5 (very poor).
Change in IC/BPS symptoms as measured by the Interstitial Cystitis Symptom Index (ICSI) | Baseline and Day 5
  The ICSI (score range: 0-19 points) and ICPI (score range: 0-16 points) contain four questions related to urinary and pain symptoms. For the ICSI, 3 of the 4 questions utilize a range of 0-5 with 0 indicating the symptom is never experienced and 5 indicating the symptom is almost always experienced. The fourth question utilizes a range of 0-4 with 0 indicating the symptom is never experienced and 4 indicating the symptom is almost always experienced.
Change in IC/BPS symptoms as measured by the Interstitial Problem Index (ICPI) | Baseline and Day 5
  For the ICPI, all four questions utilize a range of 0-4 with 0 indicating it is no problem and 4 indicating a big problem.
Change in IC/BPS symptoms as measured by the Pelvic Pain and Urgency/Frequency (PUF) Patient Symptom Scale | Baseline and Day 5
  The PUF Patient Symptom Scale is a validated instrument used to assess the severity of symptoms associated with IC/BPS and the degree to which these symptoms "bother" a patient. It is separated into 2 subsections, scored individually as the Symptom Score and Bother score, to produce one composite score. The symptom score is comprised of 7 items addressing urinary frequency, urgency, nocturia, dyspareunia, and pelvic pain. Each item is scored from 0 (never) to 3 (always) or 1 (mild) to 3 (severe), except for two which quantify daytime frequency and nocturia separately with scores ranging from 0 to 4. A composite score between 10 and 14 indicates a strong diagnosis of IC/BPS with higher scores reflecting a greater degree of severity of symptoms and disease progression as well as impact on quality of life.
Change in pelvic pain, as measured by the Brief Pain Inventory (BPI) Short Form | Baseline and Day 5
  The BPI Short Form is a validated questionnaire to assess the severity of systemic and pelvic pain and its interference in overall quality of life. Pain severity is measured through four 11-point numeric rating scales (NRS) assessing pain at its "worst," "least," and "average," within the past week, and pain "right now" (at the time of short form completion), with the composite (mean score) of all four scales indicating overall pelvic pain. Pain interference is measured through 7 scales, with scores ranging from 0 (does not interfere) to 10 (completely interferes), for different daily activities. The composite score for the interference items is used to assess overall pain interference, with higher scores indicating greater symptom severity and a change in 2 points indicating a significant change in pain. The form also consists of 3 pain body maps to identify specific locations of pain, and 2 questions related to the effect of current medications on pain.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Walker, PhD, Principal Investigator — Wake Forest University Health Sciences

IPD SHARING:
Plan to Share IPD: No